CLINICAL TRIAL: NCT05162560
Title: Incidence of Acute Diverticulitis in Finland: Nationwide Register Study of Epidemiology and Outcome of Treatment Between 2009-19
Brief Title: Incidence and Outcome of Acute Diverticulitis in Finland
Status: Recruiting | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: Tampere University Hospital (Other); Mikkeli Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 5200661
Record Dates: First submitted 2021-10-25; First posted 2021-12-17 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Acute Diverticulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patients with acute diverticulitis — registry and hospital charts of patients with acute diverticulitis

SUMMARY:
The incidence of acute diverticulitis (AD), conservative vs. surgical treatment and outcome of patients are studied using national registries and patient charts from two hospitals between years 2009-19.

DETAILED DESCRIPTION:
Acute diverticulitis (AD) of colon is increasing in Finland. Incidence, prevalence and mortality of AD of colon are investigated during 10-year period (2009-2019) in whole country. Epidemiological data is compared to data of acute appendicitis. Nationwide data of patients with AD are asked from Finnish Institute for Health and Welfare (THL). To compare registry-based nationwide data, patient charts from electronic database of two hospitals (Mikkeli Central Hospital and Tampere University Hospital) are reviewed from same study period. Patient characteristics, medication, treatment (conservative vs surgery), recurrence of AD and long-term outcome are recorded.

ELIGIBILITY:
Inclusion Criteria:

* all patients with acute diverticulitis (K57) in Finland and in two hospitals

Exclusion Criteria:

* other reasons for acute or chronic abdominal pain

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with acute diverticulitis is whole Finland and in two study hospitals during years 2009-2019
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of annual incidence and prevalence of acute diverticulitis | January 2009-December 2019
  how many patients with acute diverticulitis are treated in all hospitals in Finland

SECONDARY OUTCOMES:
Number of patients with surgical or conservative treatment | January 2009-December 2019
  Number of patients with conservative or surgical treatment of acute diverticulitis in two hospitals
Number of treatment complications and survival of patients with acute diverticulitis | January 2009-December 2019
  outcome of patients with acute diverticulitis in two hospitals

CONTACTS AND LOCATIONS:
Overall Officials: Hannu EK Paajanen, MD, Principal Investigator — Eastern Univerisity of Finland
Locations (1):
- Mikkeli Central Hospital, Mikkeli, Finland

IPD SHARING:
Plan to Share IPD: No